CLINICAL TRIAL: NCT04165980
Title: Effects of Non-invasive Brain Stimulation Methods in Experimentally Induced Pain
Brief Title: Modulatory Effects of Multichannel tDCS During Prolonged Experimental Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Luisina Gregoret, PhD Fellow, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: VN-20180092
Record Dates: First submitted 2019-11-14; First posted 2019-11-18 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Prolonged Pain; Neuroplasticity; Brain Modulation
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: The current studies have a randomized, parallel, sham-controlled and double-blinded design.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham transcranial direct current stimulation (sham tDCS) (Sham Comparator): This study has a parallel design and 2 groups: Active tDCS and Sham tDCS. Sham tDCS applies a standard sham protocol consisting of ramping up and down during 30 seconds at the beginning and at the end of each tDCS session. Each tDCS session lasts 20 minutes and applies a total current of 4mA.
  Interventions: Device: transcranial direct current stimulation
- Active transcranial direct current stimulation (activetDCS) (Active Comparator): The active comparator is the Active tDCS group. The active tDCS will target the resting-state motor network and will apply a distributed direct current during the whole session. (The TIME during the direct current is applied is the only difference with Sham tDCS) Each tDCS session lasts 20 minutes and applies a total current of 4mA.
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — Transcranial direct current stimulation delivers a low intensity current of up to 4 mA per session through small and circular shaped electrodes applied over the scalp. This induces a weak but focal electrical field that may modify the excitability of the underlying cortical target in a polarity and activity dependent fashion.

SUMMARY:
Corticomotor excitability, pain sensitivity, descending pain control and somatosensory evoked potentials (SEPs) is often altered in acute and chronic pain.

Topical capsaicin generates stable, long-lasting hyperalgesia and ongoing tonic pain in healthy participants, which significantly inhibits corticomotor excitability in the primary motor cortex (M1).

Recent studies (by Fischer et al 2017) indicated that multifocal Transcranial Direct Current Stimulation (tDCS) administered to brain regions linked to the resting state motor network (network-tDCS) could enhance corticomotor excitability in healthy participants compared to single site M1-tDCS.

It remains unknown whether network-tDCS has also the potential to modulate the inhibitory effects on motor cortex excitability, pain sensitivity, descending pain control and SEPs associated with prolonged pain

DETAILED DESCRIPTION:
To date, pain modulation to M1 rs-network tDCS during 8% capsaicin induced pain has not been assessed (Mylius, Borckardt and Lefaucheur, 2012). Further, it is unknown how multichannel tDCS acts on tonic cutaneous pain for approximately 24 hours.

The main objective of these projects are to study and characterize quantitatively the effects of multichannel tDCS in the development of prolonged pain.

It is hypothesized that multichannel tDCS of left M1 resting-state network will reduce the severity of experimentally prolonged pain over the m. first dorsal interosseous (FDI), will increase descending pain control, might possibly increase pain thresholds and simultaneously will modulate the peak-to-peak amplitude of SEPs to electrical painful stimulation. Further, it is hypothesized that descending pain modulation of M1 tDCS will be related to interference with the suppression of cortical excitability

ELIGIBILITY:
Inclusion Criteria:

-Right-handed healthy men and women in the age 21-50 years who speak and understand English

Exclusion Criteria:

* Lack of ability to cooperate
* History of chronic pain or current acute pain
* Pregnancy
* Drug addiction defined as the use of cannabis, opioids or other drugs
* Present and previous neurologic, musculoskeletal or mental illnesses
* Chili allergies (subproject 1 and 2)
* Current use of medications that may affect the trial
* Previous experience with rTMS and tDCS
* Contraindications to rTMS application (history of epilepsy, metal implants in head or jaw, etc.)
* Failure to pass the questionnaire for tDCS
* Failure to pass the "TASS questionnaire" (TASS = Transcranial Magnetic Stimulation Adult Safety Screen) (Rossi et al., 2001)

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Corticomotor excitability | 24 hours
  Corticomotor excitability is expressed as the peak-to-peak amplitude of motor evoked potentials to single-pulse transcranial magnetic stimulation. It is expected that network-tDCS will reduce corticomotor inhibition induced by tonic pain during 24 hours.

SECONDARY OUTCOMES:
Conditioned pain modulation effect | 24 hours
  Conditioned pain modulation effect is an indicator of descending inhibitory control in humans. In this study, it is performed using pressure cuff algometry. The CPM protocol consisted of a constant cuff pressure stimulation (conditioning stimulus) at 70% of the PTT (recorded for pain sensitivity assessment on that day) applied to the left leg and simultaneously one ramped cuff stimulation (test stimulus) at 1 kPa/s applied to the right leg. It is hypothesized that network-tDCS might normalize the CPM effect reduced by tonic pain during 24 hours.
Warm detection thresholds (sensitivity measure) | 24 hours
  Warm detection thresholds will be assessed using a thermode applied on the volar forearm. The thermode will start increasing the temperature from 32 C (Celsius degrees) until the participant can detect a warm sensation and will immediately press a stop button. This task will be repeted a total of 4 times.
  It is hypothesized that 2 daily treatments of active network-tDCS will not modulate this sensitivity measure during prolonged pain due to a small effect size.
Heat pain thresholds (pain sensitivity measure) | 24 hours
  Heat pain thresholds will be assessed using a thermode applied on the volar forearm. The thermode will start increasing the temperature from 32 C (Celsius degrees) until the participant can detect a temperature increment from just "a warm sensation" to an additional of either "burning" or "painful" and will immediately press a stop button. This task will be repeted a total of 3 times.
  It is hypothesized that 2 daily treatments of active network-tDCS will not modulate this pain sensitivity measure during prolonged pain due to a small effect size.
Mechanical pain thresholds (pain sensitivity measure) | 24 hours
  Mechanical pain thresholds (MPT) were assessed using seven pinprick stimulators (MRC Systems GmbH, Germany) exerting forces ranging from 8 mN to 512 mN over the distal part of the volar forearm. Starting with the lightest, each stimulator is applied in an ascending order until the participant reported a perception of sharpness or pain. If the pain threshold is not reached, the value of 1024 mN was registered. The MPT will be expressed as the geometric mean of five series of ascending/descending series of stimuli.
  It is hypothesized that 2 daily treatments of active network-tDCS will not modulate this pain sensitivity measure during prolonged pain due to a small effect size.
Cuff pressure pain sensitivity | 24 hours
  A computer-controlled cuff algometer combined with two 10-cm wide air-pressured cuffs and an electronic visual analogue scale (eVAS; anchored at 0 cm [no pain] and 10 cm [worst pain imaginable]) are used to assess cuff pressure pain detection thresholds (PDT) and pain tolerance thresholds (PTT).
  It is hypothesized that 2 daily treatments of active network-tDCS will not modulate these pain sensitivity measures during prolonged pain due to a small effect size.
Amplitude of SEPs to electrical painful stimulation | 24 hours
  It is expected that the peak to peak amplitude of SEPs (in Cz position) will be modulated by tonic pain during 24 hours and by network-tDCS.
Latency of SEPs to electrical painful stimulation | 24 hours
  it is expected that the latency of SEPs will remain unchanged during the 24 hours period and will not be affected by neither prolonged pain nor by network-tDCS.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Graven-Nielsen, PhD, Principal Investigator — Aalborg University
Locations (1):
- Aalborg University, Aalborg, Nordylland, Denmark

IPD SHARING:
Plan to Share IPD: Undecided